CLINICAL TRIAL: NCT05454488
Title: An Evidence-Based Focal Cryotherapy Protocol for Focal Ablation of Intermediate Risk Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0165; NCI-2022-05462 (Other: NCI-CTRP Clinical Trials Reporting Registry)
Record Dates: First submitted 2022-06-28; First posted 2022-07-12 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Focal therapy Treatment (Experimental): Cryoablation is a procedure in which special needles are inserted into the tumor site.
  Interventions: Drug: Focal Cryoablation; Other: Standard of Care; Other: Quality-of-life Questionnaires

INTERVENTIONS:
Drug: Focal Cryoablation — Participants will have the Focal cryoablation placed by the needles in such a way that the area of affected tissue is much smaller and focus just on the tumor tissue and surrounding area
Other: Standard of Care — Participants will receive a prostate biopsy.
Other: Quality-of-life Questionnaires — Participants will fill out questionnaires.

SUMMARY:
To learn if using cryotherapy to treat only the part of the prostate known to contain cancer is effective in controlling prostate cancer

DETAILED DESCRIPTION:
Primary Objective:

• To determine the effectiveness of an evidence-based focal cryotherapy ablation by measuring negative in-field recurrence rate at 6-months post-ablation.

Secondary Objectives:

* To determine quality of life following focal prostate cancer ablation using validated questionnaires (EPIC-26, AUA symptoms score, SHIM).
* To establish PSA kinetics post-evidence-based focal cryotherapy ablation.
* To determine rates of out of field recurrence on 6-month biopsy following focal cryotherapy ablation.
* To determine MRI findings post-focal cryotherapy ablation, including those related to prostate and surrounding periprostatic fat volume.
* To determine rate of progression and re-intervention collected as part of standard of care treatment for 5-year following study treatment.
* To describe financial toxicity associated with focal prostate cancer treatment using cryotherapy.
* To describe the incidence and severity of complications within 30-days after the study focal ablation treatment.
* To describe imaging findings on PSMA PET MRI performed in a subset of men after standard of care focal cryotherapy prior to 6-month biopsy.

ELIGIBILITY:
Inclusion criteria:

* English-speaking adult males
* Life expectancy over 10 years as assessed by treating physician
* Prior to enrollment, MRI fusion biopsy of MRI-visible lesion required (as detailed below, which includes systematic biopsy cores)
* Single focus GG2 or GG3 (additional GG1 allowed up to 6mm, noting that a single focus of disease is defined as an area seen on MRI that may be biopsied multiple times using targeted biopsies and have systematic core biopsies directly adjacent to targeted cores; all of which being considered as from the same focus)

  * Histologically confirmed adenocarcinoma of prostate
  * Organ-confined prostate cancer, clinical stage ≤T2bN0M0
  * Visible tumor on MRI
  * No clear evidence or high suspicion of extraprostatic extension or seminal vesical invasion on MRI
  * Biopsy via transperineal or transrectal approach with at least 2 cores of MRI visible lesions that are PIRADS 2 or higher and 12 core systematic biopsy template (exclusion of cores from systematic template that overlap with targeted cores allowed).
  * Additional performance of microultrasound guided biopsy is allowed though not required. Please note that every effort will be made to correlate microultrasound findings with MRI, in order to determine if positive results are from the same MRIvisible focus. This determination will be made by the surgeon performing the biopsy.
  * Note that GGG 1 disease at sites other than ablation zone are allowed provided these are 6mm or less in size. PSA ≤15 ng/mL, or PSAD <0.15 if PSA >15 ng/mL
* Physician can fully visualize the prostate on transrectal ultrasound on entry biopsy
* Lesion anatomically amenable to cryotherapy treatment based on treating physician's discretion
* Willing and able to read, understand and sign the study specific informed consent document
* Willing and agreeable to comply with study protocol requirements, including focal cryotherapy ablation and all follow up visit requirements
* Patients must consent to investigative laboratory protocol (such as, but not limited to, 2021- 0560)

Exclusion criteria:

* Gleason grade group 4 or 5 disease
* Medical history or concurrent disease, which in the opinion of the investigator, poses the patient at significant peri-operative risk of complication due to anesthesia or the procedure
* Active urinary tract infection
* Any previous treatment for prostate cancer, including radiation therapy, hormonal treatment, biologic therapy for prostate cancer, or chemotherapy
* Prior TURP or other prostate outlet procedure such as HoLEP, greenlight, microwave ablation, aquablation, UroLift, or simple prostatectomy.
* Previous rectal surgery (other than hemorrhoidectomy) or history of rectal disease
* Inability to obtain prostate MRI (ex. due to claustrophobia, pacemaker, or prohibitive implants)
* Unwilling to consent to laboratory investigative protocol (such as, but not limited to, 2021- 0560)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-07-25 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Quality-of-life Questionnaires | through completion an average of 1 year.
  Score scale ranges (0-5) 0-Not at all/5- Almost always

CONTACTS AND LOCATIONS:
Overall Officials: Justin Gregg, MD, Principal Investigator — jrgregg@mdanderson.org
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org